CLINICAL TRIAL: NCT01058486
Title: Multicomponent Intervention to Decrease COPD-related Hospitalizations
Brief Title: Multicomponent Intervention to Decrease Chronic Obstructive Pulmonary Disease (COPD)-Related Hospitalizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-004341
Record Dates: First submitted 2010-01-22; First posted 2010-01-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Disease Management; Physical Activity; Self-efficacy; Self management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Self-Management; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activity-Self Management (Experimental)
  Interventions: Behavioral: Self-Management and Motivational Interviewing
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Self-Management and Motivational Interviewing — Post hospital discharge, patients will be referred (<2 weeks) to pulmonary rehabilitation (PR) (1-2 sessions per week for 6-8 weeks). PR visits (approximately 1 hour) will include education, strengthening and endurance exercise as the patient tolerates.
  A counselor (RN or RRT) and patient will meet once weekly after PR session. The counselor will assess the patient's self efficacy and knowledge of self-management principles of COPD. Based on the assessment and greatest needs identified by patient, the counselor will work with the participant to collaboratively develop a specific SM plan.Motivational interviewing techniques will be used.
  Following completion of PR, the counselor will contact the patient monthly to provide clinical support on SM of COPD. To ensure consistency of intervention, we will use standardized treatment procedures and phone scripts.
  Arms: Activity-Self Management

SUMMARY:
The investigators' proposed study is a randomized controlled trial that will prospectively examine the effect of a multicomponent intervention on the rate of hospitalizations, daily physical activity, self efficacy and health status in patients who have COPD and have been hospitalized because of a COPD exacerbation.

In the study, a convenience sample of patients recently hospitalized for a COPD exacerbation, who meet the selection criteria and agree to participate will be randomized to receive one of the following at the time of hospital discharge: (1) the current standard of care plus a multicomponent intervention (counselor + pulmonary rehabilitation) or (2) the current standard of care without the intervention.

This study plans to test the following hypotheses: (1) The primary outcome of the study to be the composite endpoint of death or COPD hospitalization (2) Time to first rehospitalization will be shorter in the intervention group than the control group (3) At follow-up, the physical activity level measured in terms of the average number of steps and active energy expenditure will be higher in the intervention group than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥40 years old
* Clinical diagnosis of COPD or pulmonary function testing reflecting an FEV1/FVC ratio of <0.70
* Current or previous smoker with at least 10 pack-years of cigarette smoking
* Recently hospitalized for an exacerbation of COPD

Exclusion Criteria:

* Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency, are planning to move out of the state, are not living in the healthcare area, or have no telephone at home).
* Patents with characteristics that can confound the analysis of the primary outcome (patients who are living in a nursing home, have unresectable lung cancer, or have another advanced neoplasm).
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).
* Patients with an inability to do mild exercise, such as cycling or walking, when their COPD is stable (patients who have orthopedic-neurologic problems; patients who have severe heart failure, characterized by an ejection fraction of <20% or by New York Heart Association Class IV disease; patients who should be at complete rest, confined to a bed or chair; or patients in whom any physical activity brings on discomfort and in whom symptoms occur at rest).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To determine the impact of the intervention initiated after hospital discharge from a COPD exacerbation on the rate of COPD related re-hospitalizations in the intervention versus the control group . | 12 months
  "a priori" measure as funded by NIH
To determine the impact of the intervention initiated after hospital discharge from a COPD exacerbation on the rate of the composite outcome, COPD related hospitalizations or death in the intervention versus the control group. | 12 months

SECONDARY OUTCOMES:
To determine the impact of the intervention on self efficacy for physical activity and disease management, physical activity level and active energy expenditure, and health-related quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota

REFERENCES:
- [Derived] Benzo R, McEvoy C. Effect of Health Coaching Delivered by a Respiratory Therapist or Nurse on Self-Management Abilities in Severe COPD: Analysis of a Large Randomized Study. Respir Care. 2019 Sep;64(9):1065-1072. doi: 10.4187/respcare.05927. Epub 2019 Mar 26. PMID 30914491
- [Derived] Benzo R, Vickers K, Novotny PJ, Tucker S, Hoult J, Neuenfeldt P, Connett J, Lorig K, McEvoy C. Health Coaching and Chronic Obstructive Pulmonary Disease Rehospitalization. A Randomized Study. Am J Respir Crit Care Med. 2016 Sep 15;194(6):672-80. doi: 10.1164/rccm.201512-2503OC. PMID 26953637
- [Derived] Benzo R, Wetzstein M, Neuenfeldt P, McEvoy C. Implementation of physical activity programs after COPD hospitalizations: Lessons from a randomized study. Chron Respir Dis. 2015 Feb;12(1):5-10. doi: 10.1177/1479972314562208. Epub 2014 Dec 15. PMID 25511306